CLINICAL TRIAL: NCT05453240
Title: Post-Approval Study - Post-Market Surveillance Study to Evaluate the Long-Term Safety and Effectiveness of the LVIS® Device
Brief Title: Post-Market Surveillance Study to Evaluate the Long-Term Safety and Effectiveness of the LVIS Device
Acronym: LVIS PAS
Status: Enrolling by invitation | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL11008
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The proposed study is a multi-center single arm retrospective and prospective data collection, of patients treated with the LVIS device of specific sizes of 3.5mm, 4.0mm, 4.5mm, 5.5mm with up to 5 years follow-up. Information collected during the study will be standardized across centers to include pre-treatment baseline characteristics of patients including aneurysm(s) symptoms, procedural information, prespecified clinical safety events of interest, and follow-up imaging, clinical visits or telephone calls.

ELIGIBILITY:
Inclusion Criteria:

The following criteria match the FDA-approved indications for use per PMA (P170013)

* Subjects treated with the LVIS® Device in accordance with currently approved indications for use;
* Treatment of wide-necked (neck ≥ 4mm or dome to neck ratio < 2) intracranial saccular aneurysm arising from a parent vessel with a diameter ≥ 2.0 mm and ≤ 4.5 mm who underwent treatment with LVIS device of researched sizes within the last 5 years.

(Device models: 212517-LVIS, 212525-LVIS, 213015-LVIS, 213025-LVIS, 213041-LVIS, 214035-LVIS, 214049-LVIS; 212912-LVIS, 212917-LVIS, 212922-LVIS, 212928-LVIS, and 212931-LVIS);

* Availability of Medical Health Records;
* Subject whose age is ≥ 18;
* Appropriate or Waived Consent:

  1. For retrospective review: Local Institutional Review Board approves the research as exempt, allowing an all-inclusive retrospective examination of medical records documenting treatments using the study devices and available clinical and imaging follow up;
  2. For prospective follow up: Subject or his/her Legally Authorized Representative consents to participation in the study follow up visits up to 5 years, and provides a signed informed consent form as applicable;.

Exclusion Criteria:

* Subjects not treated according to the currently approved indications for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population conforms to currently approved Indications for Use: Subjects with wide-necked (neck ≥ 4 mm or dome to neck ratio < 2) intracranial, saccular aneurysms arising from a parent vessel with a diameter ≥ 2.0 mm and ≤ 4.5 mm who underwent treatment with LVIS device since approval in the local geography of researched sizes.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete or Stable Raymond Roy II | 5 year
  The Raymond-Roy occlusion classification (RROC) is an angiographic classification scheme for grading the occlusion of endovascularly treated intracranial aneurysms. It is also known as the Raymond class, Montreal scale or the Raymond Montreal scale
Intracranial hemorrhage including SAH and IPH | 5 year
  Determined by adverse event adjudication by the clinical events committee
All ischemic and hemorrhagic stroke | 5 year
  Determined by adverse event adjudication by the clinical events committee
Neurological deaths | 5 year
  Determined by adverse event adjudication by the clinical events committee
Transient Ischemic Attack | 5 year
  Determined by adverse event adjudication by the clinical events committee
Parent artery patency | 5 year
  Determined by the corelab adjudication of images
In-stent stenosis | 5 year
  Determined by the corelab adjudication of images
Target aneurysm retreatment | 5 year
  Presented by the subject medical records
Cerebral vasospasm | 5 year
  Presented by the subject medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Microvention, Aliso Viejo, California, United States